CLINICAL TRIAL: NCT06853431
Title: Determination of ED50 and ED95 With Clinical Efficacy of Intranasal Dexmedetomidine Combined With Esketamine for Preoperative Sedation in Pediatric General Anesthesia
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2025-03-105
Record Dates: First submitted 2025-02-24; First posted 2025-03-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Preoperative Anxiety; Preoperative Sedation; Children; Dexmedetomidine; Esketamine; ED95; ED50; Preoperative Sedation of Children
Keywords: Preoperative Anxiety; Preoperative sedation; Children; Dexmedetomidine; Esketamine; ED95; ED50; preoperative sedation of children
MeSH Terms: interventions — Dexmedetomidine; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1-3 years old (Experimental): The sedation depth of the children was assessed using the Ramsay Sedation Scale. This study was conducted using the biased coin design up - and - down method. The dose for the subsequent participant was determined based on the response of the previous participant. If the previous participant achieved successful sedation, the next participant had a 95% probability of receiving the same dose of dexmedetomidine as the previous participant and a 5% probability of receiving a lower dose of dexmedetomidine (a dose reduction of 0.25 µg/kg). If the previous participant failed to achieve sedation, the dose of dexmedetomidine for the next participant was increased by 0.25 µg/kg until the number of participants reached 40.
  Interventions: Drug: dexmedetomidine; Drug: Esketamine
- 3-6 years old (Experimental): The sedation depth of the children was assessed using the Ramsay Sedation Scale. This study was conducted using the biased coin design up - and - down method. The dose for the subsequent participant was determined based on the response of the previous participant. If the previous participant achieved successful sedation, the next participant had a 95% probability of receiving the same dose of dexmedetomidine as the previous participant and a 5% probability of receiving a lower dose of dexmedetomidine (a dose reduction of 0.25 µg/kg). If the previous participant failed to achieve sedation, the dose of dexmedetomidine for the next participant was increased by 0.25 µg/kg until the number of participants reached 40.
  Interventions: Drug: dexmedetomidine; Drug: Esketamine

INTERVENTIONS:
Drug: dexmedetomidine — esketamine 0.5mg/kg intranasally via a nasal dropper, dexmedetomidine 1μg/kg was given intranasally, and the adjusted dose of dexmedetomidine was 0.25μg/kg.
Drug: Esketamine — esketamine 0.5mg/kg intranasally via a nasal dropper, dexmedetomidine 1μg/kg was given intranasally, and the adjusted dose of dexmedetomidine was 0.25μg/kg.

SUMMARY:
For pediatric patients undergoing general anesthesia, poor anesthesia induction compliance often has adverse effects on individual behavior in the early postoperative period. Dexmedetomidine can reduce the cardiovascular responses and postoperative mental adverse reactions caused by esketamine anesthesia induction [6]. This study aims to explore the ED50 and ED95 and clinical effects of the combination of dexmedetomidine and esketamine nasal drops for preoperative sedation in children of different ages undergoing general anesthesia, providing a theoretical basis for the combined use of dexmedetomidine and esketamine for preoperative sedation in children undergoing general anesthesia.

DETAILED DESCRIPTION:
Children scheduled for general anesthesia were randomly divided into two groups based on age: Group T consisted of toddlers aged 1 - 3 years old, and Group P consisted of preschool children aged 3 - 6 years old. The initial dose for both groups was dexmedetomidine 1μg/kg and esketamine 0.5mg/kg.

The sedation depth of the children was assessed using the Ramsay Sedation Scale. An unbiased coin - flipping design was adopted: after esketamine 0.5mg/kg was administered intranasally via a nasal dropper, dexmedetomidine 1μg/kg was given intranasally. The adjusted dose of dexmedetomidine was 0.25μg/kg. If the sedation of the previous child failed, the intranasal dose of dexmedetomidine for the next child would be increased by 0.25μg/kg. If the sedation of the previous child was successful, a card would be drawn to decide the induction dose for the next patient. A total of 20 cards, which were identical in appearance, were prepared. The probability of administering the same dose was 19/20 (95%), and the probability of reducing the dose for the next patient by 0.25μg/kg was 1/20 (5%).

After drug administration, an anesthesiologist who was unaware of the medication usage would rate the sedation level using the Ramsay Sedation Scale every 5 minutes. The non - invasive blood pressure (NIBP), heart rate (HR), respiratory rate (RR), and blood oxygen saturation (SpO2) were recorded before drug administration (0 minutes, baseline) and at 5, 10, 15, 20, 25, and 30 minutes after drug administration.The onset time was defined as the time from intranasal administration to an RSS score of ≥ 4. Thirty minutes after intranasal administration, an experienced nurse who was unaware of the intranasal drug dose performed intravenous cannulation. The emotional state was assessed using the Emotional State Scale (ESS - 4) during intravenous cannulation. Successful intravenous cannulation was defined as an ESS - 4 score of ≤ 2 during cannulation, regardless of whether the intravenous infusion catheter was successfully inserted.The Pediatric Anesthesia Emergence Delirium (PAED) scale was used to assess the degree of emergence delirium in children. The onset time of sedation (the time to reach an RSS score of ≥4 after intranasal drug administration), surgical time (from the start to the end of the surgery), and awakening time (from the closure of the sevoflurane vaporizer to an Aldrete score of 9 or above) were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status classification Grade I or II;
2. Age 1-6 years old;
3. Children who need to undergo general anesthesia for elective surgery;
4. Weight within the normal range;
5. Signed informed consent form. -

Exclusion Criteria:

1. The child's guardian or the child themselves refuses to participate in the study;
2. Patients with contraindications for sedation/anesthesia or a history of abnormal recovery from sedation/anesthesia;
3. Individuals known to be allergic to the study drugs, opioid drugs, or rescue medications;
4. Individuals with a history of heart, brain, liver, kidney, or metabolic diseases;
5. Individuals with an upper respiratory tract infection within the past two weeks;
6. Individuals with other diseases that may cause harm to the subject. -

Ages: 12 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Onset time of sedation | Within 30 minutes after intranasal administration of dexmedetomidine.
  After drug administration, every 5 minutes, an anesthesiologist who was unaware of the medication used assessed the sedation level using the Ramsay Sedation Scale(RSS).Within 30 minutes after the intranasal medication was administered, the Ramsay Sedation Score (RSS) was ≥4.

SECONDARY OUTCOMES:
Intravenous cannulation success rates | 30 minutes after intranasal administration of dexmedetomidine.
  Emotional State Score
  1. Calm
  2. Apprehensive, not smiling, tentative behavior, withdrawn
  3. Crying
  4. Thrashing, crying with movements of the arms and legs, resisting
Awakening time | Within 1 hour of entering the Post Anesthesia Care Unit (PACU).
  From the closure of the sevoflurane vaporizer to the time when the patient opened their eyes.
Postoperative agitation | Within up to 15-30 minutes after child's first eye opening in the postoperative period
  The pediatric anesthesia emergence delirium scale consists of five items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score. pediatric anesthesia emergence delirium scale ≥12 at any time indicates presence of emergence delirium.
Number of children with adverse effects | Up to 24 hours including preoperative, intraoperative, and postoperative periods
  １、Bradycardia and/or hypotension need for hemodynamic support; 2、Desaturation is defined as Oxygen desaturation <90%; 3、Nausea and vomiting; 4、Any adverse effects requiring interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No